CLINICAL TRIAL: NCT04193878
Title: ARrest RESpiraTory Failure From PNEUMONIA (ARREST PNEUMONIA)
Brief Title: ARrest RESpiraTory Failure From PNEUMONIA
Acronym: ARREST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per DSMB's review of interim analysis, the study has reached the pre-specified futility criteria
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Joseph Levitt, MD, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 53599; 1UG3HL141722-01A1 (NIH)
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Pneumonia; Hypoxemia; Acute Respiratory Failure; COVID-19 Pneumonia
MeSH Terms: conditions — Pneumonia; Hypoxia | interventions — Formoterol Fumarate; Budesonide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 4 ml aerosolized 0.9% saline every 12 hours x 10 doses
  Interventions: Drug: Inhaled placebo
- Intervention (Active Comparator): aerosolized formoterol (20 mcg/2 ml) and budesonide (1.0 mg/2 ml) every 12 hours x 10 doses
  Interventions: Drug: Inhaled budesonide and formoterol

INTERVENTIONS:
Drug: Inhaled budesonide and formoterol — aerosolized doses of budesonide (1.0 mg/2 ml) and formoterol (20 mg/2 ml) twice daily for up to 5 days
  Other Names: Pulmicort Respules (budesonide) and Perforomist (formoterol)
  Arms: Intervention
Drug: Inhaled placebo — aerosolized saline (4 ml of 0.9% saline) twice daily for up to 5 days
  Other Names: aerosolized 0.9% saline
  Arms: Placebo

SUMMARY:
This research study seeks to establish the effectiveness of a combination of an inhaled corticosteroid and a beta agonist compared to placebo for the prevention of acute respiratory failure (ARF) in hospitalized patients with pneumonia and hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years or older with

Severe pneumonia defined as:

1. Hospitalization for acute (defined as ≤ 14 days) onset of symptoms (cough, sputum production, or dyspnea), AND 2. Radiographic evidence of pneumonia by chest radiograph or CT scan, AND 3. One of the following:

1. Evidence of systemic inflammation (temperature < 35◦C or > 38◦C OR WBC > or < upper or lower limits for site OR procalcitonin > 0.5 mcg/L), OR
2. Known current immunosuppression preventing inflammatory response, OR
3. High clinical suspicion of pneumonia with microbiologic confirmation of infection. Microbiologic confirmation will include a positive nasal swab for a known respiratory virus; a sputum culture growing a likely pathogenic organism plus moderate or greater WBCs (not required for immunocompromised patients); or a positive blood culture with a likely pathogenic organism - e.g., ¼ vials with S. Epidermidis would NOT qualify)

AND Hypoxemia defined as new requirement for daytime supplemental oxygen with SpO2 < 92% on room air, ≤ 96% on ≥ 2 L/min oxygen, or > 6L/min or non-invasive ventilation regardless of SpO2 at enrollment. Patients admitted with pneumonia but not meeting criteria for hypoxemia will be followed for up to 48 hours from ED admission to enrolling hospital to assess for development of qualifying hypoxemia.

Exclusion Criteria:

* Inability to randomize within 48 hours of presentation to enrolling hospital (randomization beyond 24 hours will be limited to patients with persistent hypoxemia defined by an SpO2 < 97% while on > 3L/min O2)
* Intubation (or impending intubation) prior to enrollment

  a. Patients receiving HFNC oxygen or NIV prior to enrollment are not excluded
* A condition requiring inhaled corticosteroids or beta-agonists (patients receiving inhaled beta-agonists in the ED without an established indication will be eligible if treating clinician is willing to discontinue subsequent treatments)
* Chronic systemic steroid therapy equivalent to >10 mg prednisone
* COVID-19 positive patients receiving > 6 mg dexamethasone (40 mg prednisone equivalent dose) except for stress dose steroids for septic shock
* Non-COVID-19 pneumonia patients receiving systemic steroid > 10 mg prednisone except for stress dose steroids for septic shock
* Chronic lung or neuromuscular disease requiring daytime oxygen or mechanical ventilation other than for obstructive sleep apnea (OSA) or obesity hypoventilation syndrome
* Not anticipated to survive > 48 hours or not expected to require > 48 hours of hospitalization
* Contraindication or allergy to inhaled corticosteroids or beta-agonists
* Patients with heart rate > 130 bpm, ventricular tachycardia or new supraventricular tachycardia within last 4 hours will be potentially eligible for enrollment after the condition has resolved
* Patients with K+ < 3.0 will be potentially eligible for enrollment after the condition has resolved
* Patient not committed to full support other than intubation or resuscitation (i.e., DNR/DNI status allowed)
* Pregnancy
* Incarcerated individual
* Physician refusal of consent to protocol
* Patient/surrogate refusal of consent to protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Acute respiratory failure (ARF) | within 7 days of randomization
  High flow nasal cannula (HFNC >=20L/mon O2) and/or Noninvasive ventilation (NIV) use for greater than 36 hours OR Invasive mechanical ventilation for greater than 36 hours OR Death in a patient placed on respiratory support (HFNC, NIV, ventilator) who dies before 36 hours

SECONDARY OUTCOMES:
Hospital length of stay | within 60 days of randomization
Duration of need for supplemental oxygen | within 30 days of randomization
Proportion of patients intubated for respiratory failure | Within 7 days of randomization
Oxygen failure free days to day 28 | Until Day 28
Progression to systemic steroid therapy for pneumonia | during course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Levitt, MD, Principal Investigator — Stanford University; Emir Festic, MD, Principal Investigator — Mayo Clinic
Locations (12):
- United States (12):
  - University of Alabama Birmingham - Main & Highlands, Birmingham, Alabama
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - University of Arizona - Main & South Campus, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - University of Florida, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Tulane University - Main & BUMC, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University - Main Campus & Bayview, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - New York University - Langone Health, New York, New York
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levitt JE, Festic E, Desai M, Hedlin H, Mahaffey KW, Rogers AJ, Gajic O, Matthay MA; ARREST Pneumonia Clinical Trial Investigators. The ARREST Pneumonia Clinical Trial. Rationale and Design. Ann Am Thorac Soc. 2021 Apr;18(4):698-708. doi: 10.1513/AnnalsATS.202009-1115SD. PMID 33493423
- [Derived] Nicolau DV, Bafadhel M. Inhaled corticosteroids in virus pandemics: a treatment for COVID-19? Lancet Respir Med. 2020 Sep;8(9):846-847. doi: 10.1016/S2213-2600(20)30314-3. Epub 2020 Jul 30. No abstract available. PMID 32738928